CLINICAL TRIAL: NCT00970632
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Global Multicenter Study to Evaluate the Efficacy and Safety of Tadalafil Once Daily Dosing for 12 Weeks in Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: A Study of Tadalafil in Men With Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12932; H6D-MC-LVID (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2011-12-23 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo tablet with tamsulosin dose orally (po) once daily (QD) and placebo capsule with tadalafil dose po QD for 12 weeks
  Interventions: Drug: Placebo tablet; Drug: Placebo capsule
- Tadalafil 5 milligram (mg) (Experimental): Tadalafil 5 mg tablet po QD and placebo capsule po QD for 12 weeks
  Interventions: Drug: Tadalafil 5 mg
- Tamsulosin 0.4 mg (Active Comparator): Tamsulosin 0.4 mg capsule po QD and placebo tablet po QD for 12 weeks
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tadalafil 5 mg — Tadalafil 5 mg po QD for 12 weeks
  Other Names: Cialis; LY450190
  Arms: Tadalafil 5 milligram (mg)
Drug: Placebo tablet — Placebo tablet po QD for 12 weeks
  Arms: Placebo
Drug: Tamsulosin — Tamsulosin 0.4 mg po QD for 12 weeks
  Arms: Tamsulosin 0.4 mg
Drug: Placebo capsule — Placebo capsule po QD for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether an experimental drug known as tadalafil given once daily can reduce the symptoms associated with Benign Prostatic Hyperplasia (straining, urinary frequency, feeling like your bladder is still full etc.)

ELIGIBILITY:
Inclusion Criteria:

* Men 45 years of age or older with benign prostatic hyperplasia (BPH) also referred to as BPH-lower urinary tract symptoms (LUTS) on the disease diagnostic criteria at the start of study.
* Provide signed informed consent at the start of the study.
* Agree not to use any other approved or experimental pharmacologic BPH, overactive bladder (OAB), or erectile dysfunction (ED) treatments anytime during the study.
* Have not taken finasteride therapy for at least 3 months before study drug is dispensed and dutasteride therapy for at least 6 months before study drug is dispensed.
* Have not taken other BPH therapy (including herbal preparations), OAB therapy, ED therapy for at least 4 weeks prior to study drug is dispensed.
* Have LUTS with a total International Prostate Symptom Score (IPSS) greater than or equal to 13 when study drug is dispensed.
* Have reduced urine flow (measured by special toilet equipment).
* Demonstrate compliance with study drug administration requirements.

Exclusion Criteria:

* Treated with nitrates
* Have unstable angina or angina that requires treatment.
* Have had any of the following in the past 90 days: Heart attack, also known as a myocardial infarction (MI); Heart bypass surgery (called coronary artery bypass graft surgery); Had a procedure to open up blood vessels in the heart known as angioplasty or stent placement (percutaneous coronary intervention).
* Have very high or very low blood pressure.
* Have certain neurological conditions associated with bladder problems or injuries to brain or spinal cord within a specified time of starting this study.
* Have uncontrolled diabetes.
* Have prostate cancer, are being treated for cancer.
* Have prostate specific antigen (PSA) greater than 10 nanograms per milliliter (ng/mL) at the start of study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (44):
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bentleigh East, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bunbury, Western Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salzburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garches
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pierre-Bénite
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suresnes
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Rappenau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Wiessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mühlacker
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oranienburg
- Greece (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ioannina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Larissa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cagliari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sassari
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saltillo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zapopan
- Netherlands (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., 's-Hertogenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arnhem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tilburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veldhoven
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kutno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw

REFERENCES:
- [Derived] Vlachopoulos C, Oelke M, Maggi M, Mulhall JP, Rosenberg MT, Brock GB, Esler A, Buttner H. Impact of cardiovascular risk factors and related comorbid conditions and medical therapy reported at baseline on the treatment response to tadalafil 5 mg once-daily in men with lower urinary tract symptoms associated with benign prostatic hyperplasia: an integrated analysis of four randomised, double-blind, placebo-controlled, clinical trials. Int J Clin Pract. 2015 Dec;69(12):1496-507. doi: 10.1111/ijcp.12722. Epub 2015 Aug 24. PMID 26299520
- [Derived] Giuliano F, Oelke M, Jungwirth A, Hatzimouratidis K, Watts S, Cox D, Viktrup L. Tadalafil once daily improves ejaculatory function, erectile function, and sexual satisfaction in men with lower urinary tract symptoms suggestive of benign prostatic hyperplasia and erectile dysfunction: results from a randomized, placebo- and tamsulosin-controlled, 12-week double-blind study. J Sex Med. 2013 Mar;10(3):857-65. doi: 10.1111/jsm.12039. Epub 2013 Jan 24. PMID 23346990
- [Derived] Oelke M, Giuliano F, Mirone V, Xu L, Cox D, Viktrup L. Monotherapy with tadalafil or tamsulosin similarly improved lower urinary tract symptoms suggestive of benign prostatic hyperplasia in an international, randomised, parallel, placebo-controlled clinical trial. Eur Urol. 2012 May;61(5):917-25. doi: 10.1016/j.eururo.2012.01.013. Epub 2012 Jan 20. PMID 22297243

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period 1: Screening and 4-week washout of benign prostatic hyperplasia (BPH), overactive bladder (OAB), and/or erectile dysfunction (ED) treatments. Period 2: 4-week, single-blind, placebo lead-in to assess compliance and establish baseline levels. Period 3: Randomization to treatment (placebo, tadalafil 5 mg, or tamsulosin 0.4 mg for 12 weeks).
Groups:
- Placebo: Placebo tablet orally (po) once daily (QD) and placebo capsule po QD for 12 weeks
- Tadalafil 5 mg: Tadalafil 5 milligram (mg) tablet po QD and placebo capsule po QD for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Started | 172 | 171 | 168
Completed | 148 | 156 | 150
Not Completed | 24 | 15 | 18
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 2
Not completed — Protocol Violation | 8 | 5 | 8
Not completed — Withdrawal by Subject | 7 | 6 | 4
Not completed — Entry criteria not met | 0 | 2 | 2
Not completed — Sponsor decision | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg | Total
Number analyzed (Participants) | 172 | 171 | 168 | 511
Age Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.65) | 63.5 (8.08) | 63.5 (7.76) | 63.6 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 172 | 171 | 168 | 511
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 47 | 43 | 139
  Not Hispanic or Latino | 123 | 124 | 125 | 372
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 41 | 40 | 37 | 118
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 131 | 130 | 131 | 392
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 6 | 9 | 10 | 25
  Austria | 13 | 10 | 7 | 30
  Belgium | 5 | 6 | 7 | 18
  France | 9 | 9 | 12 | 30
  Germany | 56 | 50 | 56 | 162
  Greece | 8 | 4 | 7 | 19
  Italy | 18 | 26 | 15 | 59
  Mexico | 43 | 41 | 38 | 122
  Netherlands | 2 | 3 | 6 | 11
  Poland | 12 | 13 | 10 | 35
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI measured the participant's body weight divided by the square of his or her height.
  kilogram per square meter (kg/m^2) | 28.1 (4.09) | 27.1 (4.03) | 27.9 (3.73) | 27.7 (3.96)
Lower Urinary Tract Symptom (LUTS) Severity [Number; unit: participants] — The total International Prostate Symptom Score (IPSS) was obtained by combining the scores of the responses to Component Questions 1-7. Each question was scored from 0-5 for a total IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represented greater severity of symptoms.
  participants
    Moderate (IPSS <20) | 118 | 123 | 119 | 360
    Severe (IPSS ≥20) | 54 | 48 | 49 | 151
Peak Urine Flow Rate (Qmax) Category [Number; unit: participants] — Qmax is a uroflowmetry parameter used to measure peak urine flow rate with a standard calibrated flowmeter in milliliters per second (mL/sec) at Visit 3 (Week 0). Percentages were based on the prevoid number of randomized participants with valid uroflowmetry data (N=498 participants). The uroflowmetry assessment was considered valid and data were included in this summary only if total bladder volume (assessed by ultrasound) was ≥150 to ≤550 mL and voided volume (V-Comp) was ≥125 mL.
  participants
    <10 mL/sec | 79 | 92 | 105 | 276
    10-15 mL/sec | 69 | 63 | 53 | 185
    >15 mL/sec | 18 | 12 | 7 | 37
Postvoid Residual Volume (PVR) [Mean (Standard Deviation); unit: milliliter (mL)] — PVR was determined by ultrasound at baseline. Urine volume was measured after complete emptying of the participant's bladder.
  milliliter (mL) | 50.9 (51.14) | 54.6 (52.29) | 59.8 (57.99) | 55.1 (53.88)
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)] — PSA is a protein produced by the cells of the prostate gland. PSA is present in small quantities in the serum of men with healthy prostates, but is often elevated in the presence of prostate disorders, such as prostate cancer.
  nanograms per milliliter (ng/mL) | 2.0 (1.69) | 2.1 (1.83) | 1.9 (1.57) | 2.0 (1.70)
Erectile Dysfunction (ED) [Number; unit: participants] — ED was defined as a consistent change in the quality of erection adversely affecting participant satisfaction with sexual intercourse.
  participants
    Yes | 120 | 121 | 116 | 357
    No | 52 | 50 | 52 | 154
Erectile Dysfunction (ED) Severity [Number; unit: participants] — ED was defined as a consistent change in the quality of erection adversely affecting subject satisfaction with sexual intercourse. Severity was based on investigator opinion. The participant population included 357 randomized subjects with ED.
  participants
    Mild | 36 | 38 | 33 | 107
    Moderate | 64 | 65 | 60 | 189
    Severe | 20 | 18 | 23 | 61
Erectile Dysfunction (ED) Duration [Number; unit: participants] — ED was defined as a consistent change in the quality of erection adversely affecting subject satisfaction with sexual intercourse. The participant population included 357 randomized subjects with ED.
  participants
    <1 year | 15 | 28 | 29 | 72
    ≥1 year | 105 | 93 | 87 | 285
Sexually Active with a Female Partner [Number; unit: participants]
  Yes | 145 | 143 | 139 | 427
  No | 27 | 28 | 29 | 84
Expect to Remain Sexually Active [Number; unit: participants] — The participant population was based on 427 randomized subjects who reported being sexually active with a female partner.
  participants
    Yes | 145 | 142 | 139 | 426
    No | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total International Prostate Symptom Score (IPSS) at 12 Weeks
Description: The IPSS Total Score was obtained by combining the scores of the responses to Component Questions 1-7. Each question was scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represented greater severity of symptoms. Least Squares (LS) Mean of change from baseline to endpoint (Week 12 or last post-baseline value carried forward) was from an analysis of covariance (ANCOVA) and adjusted for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction, and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: The analysis population included all participants who were randomized, started study medication, and had non-missing data at baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 172 | 171 | 165
units on a scale | -4.2 (0.5) | -6.3 (0.5) | -5.7 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.001, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 12 endpoint between tadalafil and placebo treatment groups was for the primary comparison and assessed for significance at a level of 0.05; Difference in LS Means = -2.1
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.023, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 12 between tamsulosin and placebo treatment groups was secondary in nature and assessed for significance at a level of 0.05 with no adjustments for multiplicity; Difference in LS Means = -1.5

2. Secondary Outcome: Change From Baseline in Total International Prostate Symptom Score (IPSS) at 4 Weeks
Description: The IPSS Total Score was obtained by combining the scores of the responses to Component Questions 1-7. Each question was scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represented greater severity of symptoms. Least Squares (LS) Mean of change from baseline to endpoint (Week 4 or last post-baseline value carried forward) was from an analysis of covariance (ANCOVA) and adjusted for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction, and treatment-by-region interaction.
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 166 | 167 | 159
units on a scale | -3.3 (0.4) | -5.5 (0.4) | -5.7 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 4 between tadalafil and placebo treatment groups was assessed for significance at a level of 0.05; Difference in LS Means = -2.2
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 4 between tamsulosin and placebo treatment groups was assessed for significance at a level of 0.05 with no adjustments for multiplicity; Difference in LS Means = -2.3

3. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Storage (Irritative) Subscore at 12 Weeks
Description: IPSS storage (irritative) subscore was the sum of Component Questions 2, 4 and 7 of the IPSS questionnaire. Scores ranged from 0 (no irritative symptoms) to 5 (frequent irritative symptoms); therefore, the 3 questions of the irritative subscore ranged from 0 to 15. Least Squares (LS) Mean of change from baseline to endpoint (Week 12 or last post-baseline value carried forward) was from an analysis of covariance (ANCOVA) and adjusted for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction, and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 172 | 171 | 165
units on a scale | -1.6 (0.2) | -2.2 (0.2) | -2.2 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.055, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 12 between tadalafil versus placebo treatment groups was assessed for significance at a level of 0.05 with no adjustments for multiplicity; Difference in LS Means = -0.6
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.055, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 12 between tamsulosin versus placebo treatment groups was assessed for significance at a level of 0.05 with no adjustments for multiplicity; Difference in LS Means = -0.6

4. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Voiding (Obstructive) Subscore at 12 Weeks.
Description: IPSS voiding (obstructive) subscore was the sum of Component Questions 1, 3, 5 and 6 of the IPSS questionnaire. Scores ranged from 0 (no obstructive symptoms)-5 (frequent obstructive symptoms); therefore, the 4 questions of the obstructive score ranged from 0-20. Least Squares (LS) Mean of change from baseline to endpoint (Week 12 or last post-baseline value carried forward) was from an analysis of covariance (ANCOVA) and adjusted for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction, and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 172 | 171 | 165
units on a scale | -2.6 (0.3) | -4.1 (0.3) | -3.5 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Difference in LS Means = -1.5
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.026, ANCOVA — [p-value comment as in outcome 3, analysis 2]; Difference in LS Means = -1.0

5. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Nocturia Question at 12 Weeks
Description: The IPSS nocturia question (Component Question 7) measured nocturia (need to urinate at night) over the past 4 weeks. Scores ranged from 0 (no episodes of nocturia)-5 (5 or more episodes of nocturia). Least Squares (LS) Mean of change from baseline to endpoint (Week 12 or last post-baseline value carried forward) was from an analysis of covariance (ANCOVA) and adjusted for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction, and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 172 | 171 | 165
units on a scale | -0.3 (0.1) | -0.5 (0.1) | -0.5 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.080, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Difference in LS Means = -0.2
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.118, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Difference in LS Means = -0.2

6. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Quality of Life (QoL) Index at 12 Weeks
Description: IPSS QoL assessed QoL by urinary symptoms, with scores ranging from 0 (delighted)-6 (terrible). Least Squares (LS) Mean of change from baseline to endpoint (Week 12 or last post-baseline value carried forward) was from an analysis of covariance (ANCOVA) and adjusted for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction, and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 172 | 171 | 165
units on a scale | -1.0 (0.1) | -1.3 (0.1) | -1.1 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.022, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Difference in LS Means = -0.3
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.546, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 12 endpoint between tamsulosin versus placebo treatment groups was assessed for significance at a level of 0.05 with no adjustments for multiplicity; Difference in LS Means = -0.1

7. Secondary Outcome: Change From Baseline in Modified International Prostate Symptom Score (mIPSS) at 1 Week
Description: The mIPSS Total Score covered a time period of 1 week and was obtained by combining scores of responses to Component Questions 1-7. Each question was scored from 0-5 for an mIPSS range of 0-35 points; higher numerical scores represented greater severity of symptoms. Least Squares (LS) Mean of change from baseline to endpoint (Week 1 or last post-baseline value carried forward) was from an analysis of covariance (ANCOVA) and adjusted for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction, and treatment-by-region interaction.
Time Frame: Baseline, 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 154 | 162 | 152
units on a scale | -2.5 (0.4) | -4.0 (0.4) | -4.0 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.003, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 1 between tadalafil and placebo treatment groups was assessed for significance at a level of 0.05; Difference in LS Means = -1.5
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.005, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 1 between tamsulosin and placebo treatment groups was assessed for significance at a level of 0.05 with no adjustments for multiplicity; Difference in LS Means = -1.5

8. Secondary Outcome: Change From Baseline in Benign Prostatic Hyperplasia Impact Index (BII) at 4 Weeks
Description: BII was a 4-item, self-administered questionnaire evaluating impact of urinary problems on overall health and activity. Total scores ranged from 0-13; higher scores represented increased perceived impact of BPH-lower urinary tract symptoms (LUTS) on overall health. Least Squares (LS) Mean of change from baseline to endpoint (Week 4 or last post-baseline value carried forward) was from an analysis of covariance (ANCOVA) and adjusted for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction, and treatment-by-region interaction.
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 166 | 167 | 159
units on a scale | -0.4 (0.2) | -1.2 (0.2) | -1.3 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Difference in LS Means = -0.8
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = -0.9

9. Secondary Outcome: Change From Baseline in Benign Prostatic Hyperplasia Impact Index (BII) at 12 Weeks
Description: BII was a 4-item, self-administered questionnaire evaluating impact of urinary problems on overall health and activity. Total scores ranged from 0-13; higher scores represented increased perceived impact of BPH-lower urinary tract symptoms (LUTS) on overall health. Least Squares (LS) Mean of change from baseline to endpoint (Week 12 or last post-baseline value carried forward) was from an analysis of covariance (ANCOVA) and adjusted for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction, and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 167 | 168 | 160
units on a scale | -0.9 (0.2) | -1.7 (0.2) | -1.5 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.003, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 12 between tadalafil and placebo treatment groups was assessed for significance at a level of 0.05; Difference in LS Means = -0.8
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.026, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 12 endpoint between tamsulosin and placebo treatment groups was assessed for significance at a level of 0.05 with no adjustments for multiplicity; Difference in LS Means = -0.6

10. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) at 12 Weeks
Description: The PGI-I was a participant-rated instrument that measured the improvement or worsening of the participant's symptoms based on a 7-point scale at Week 12. A score of 1=participant felt symptoms were "very much better"; score of 2=participant felt symptoms were "much better"; score of 3=participant felt symptoms were "a little better"; score of 4=participant felt "no change" in symptoms; score of 5=participant felt symptoms were "a little worse"; score of 6=participant felt symptoms were "much worse"; score of 7=participant felt symptoms were "very much worse".
Time Frame: 12 weeks
Population: The analysis population included all participants who were randomized, started study medication, and had non-missing data.
Measure: Number; unit: participants
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 159 | 160 | 157
participants
  Very much worse | 2 | 0 | 0
  Much worse | 2 | 1 | 0
  A little worse | 4 | 6 | 8
  No change | 51 | 28 | 36
  A little better | 53 | 52 | 55
  Much better | 36 | 56 | 48
  Very much better | 11 | 17 | 10
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — The p-value associated with difference between tadalafil versus placebo treatment groups within the 7 response categories was assessed for significance at a level of 0.05 with no adjustment for multiplicity; Analysis used data only from these treatment arms and stratification of baseline LUTS severity (moderate [total IPSS <20]; severe [total IPSS ≥20])
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.114, Cochran-Mantel-Haenszel — The p-value associated with difference between tamsulosin versus placebo treatment groups within the 7 response categories was assessed for significance at a level of 0.05 with no adjustment for multiplicity; [statistical method as in outcome 10, analysis 1]

11. Secondary Outcome: Clinician Global Impression of Improvement (CGI-I) at 12 Weeks
Description: The CGI-I was an investigator-rated instrument that measured improvement or worsening of the participant's symptoms based on a 7-point scale. A score of 1=participant felt symptoms were "very much better"; score of 2=participant felt symptoms were "much better"; score of 3=participant felt symptoms were "a little better"; score of 4=participant felt "no change" in symptoms; score of 5=participant felt symptoms were "a little worse"; score of 6=participant felt symptoms were "much worse"; score of 7=participant felt symptoms were "very much worse".
Time Frame: 12 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 160 | 163 | 157
participants
  Very much worse | 1 | 0 | 0
  Much worse | 2 | 2 | 1
  A little worse | 6 | 5 | 7
  No change | 51 | 32 | 40
  A little better | 57 | 58 | 65
  Much better | 34 | 50 | 38
  Very much better | 9 | 16 | 6
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Analysis used data only from these treatment arms and a stratification of baseline LUTS severity (moderate [total IPSS <20]; severe [total IPSS ≥20])
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.452, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 2]; [statistical method as in outcome 10, analysis 1]

12. Secondary Outcome: Treatment Satisfaction Scale - Benign Prostatic Hyperplasia (TSS-BPH) at 12 Weeks: Overall
Description: The TSS-BPH was a validated participant-rated instrument that measured participant satisfaction with treatment based on a 13-item questionnaire. The overall TSS-BPH score was converted to a percentage of the maximum value possible (percent ranged from 0-100) with lower scores indicating greater satisfaction.
Time Frame: 12 weeks
Population: The analysis population included all participants who were randomized, started study medication, and had non-missing data at baseline and at least one post-baseline measurement.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 158 | 163 | 156
units on a scale | 28.9 (17.50) | 22.2 (17.74) | 28.9 (16.49)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.005, Van Elteren Tests — The p-value associated with the testing for differences in medians between tadalafil versus placebo treatment groups was assessed for significance at a level of 0.05 with no adjustment for multiplicity; P-values testing for differences of medians between placebo and active treatment were based on the Van Elteren test, stratifying by region; Median of Treatment Group Differences = -4.4
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.457, Van Elteren Tests — The p-value associated with the testing for differences in medians between tamsulosin versus placebo treatment groups was assessed for significance at a level of 0.05 without adjustments for multiplicity; [statistical method as in outcome 12, analysis 1]; Median of Treatment Group Differences = -2.2

13. Secondary Outcome: Change From Baseline in International Index of Erectile Function (IIEF) Erectile Function (EF) Domain at 12 Weeks
Description: IIEF measured self-reported EF over the past 4 weeks. Scores ranged from 0 (low or no EF)-5 (high EF) on 6 questions (1-5, 15 of the IIEF). Total EF Domain scores ranged from 1-30. Least Squares (LS) Mean of change from baseline to endpoint (Week 12 or last post-baseline value carried forward) was from an analysis of covariance (ANCOVA) and adjusted for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction, and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: The analysis population included all randomized sexually active participants with erectile dysfunction who started study medication, and had baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 100 | 103 | 93
units on a scale | 2.1 (0.8) | 6.0 (0.8) | 1.7 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 12 between tadalafil versus placebo treatment groups was assessed for significance at a level of 0.05 with no adjustment for multiplicity; Difference in LS Means = 4.0
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.699, ANCOVA — The p-value associated with LS Mean difference of changes from baseline to Week 12 between tamsulosin versus placebo treatment groups was assessed for significance at a level of 0.05 with no adjustment for multiplicity; Difference in LS Means = -0.4

14. Secondary Outcome: Change From Baseline in Peak Urine Flow Rate (Q-Max) at 12 Weeks
Description: Q-max (peak urine flow rate) was measured in milliliters per second (mL/sec) using a standard calibrated flowmeter. At each visit, a uroflowmetry assessment was considered valid and data were included in the analyses only if the prevoid total bladder volume (assessed by ultrasound) was ≥150 to ≤550 mL and the voided volume (V-comp) was ≥125 mL.
Time Frame: Baseline, 12 weeks
Population: The analysis population included all randomized participants who started study medication, and had non-missing data at baseline and at endpoint (last non-missing post-baseline value).
Measure: Median (Standard Deviation); unit: milliliters per second (mL/sec)
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 147 | 156 | 144
milliliters per second (mL/sec) | 0.3 (4.84) [-1.5 to 3.1] | 1.6 (5.49) [-0.7 to 5.2] | 1.6 (4.06) [-0.6 to 4.1]
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.009, ANOVA — The p-value associated with median difference of changes from baseline to Week 12 endpoint between tadalafil versus placebo treatment groups was assessed for significance at a level of 0.05 with no adjustment for multiplicity; Analysis of variance (ANOVA) using rank transformed data
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.014, ANOVA — The p-value associated with median difference of changes from baseline to Week 12 endpoint between tamsulosin versus placebo treatment groups was assessed for significance at a level of 0.05 with no adjustment for multiplicity; ANOVA using rank transformed data

15. Secondary Outcome: Change From Baseline in Mean Urine Flow Rate (Q-Mean) at 12 Weeks
Description: Q-mean (mean urine flow rate) was measured in milliliters per second (mL/sec) using a standard calibrated flowmeter. At each visit, a uroflowmetry assessment was considered valid and data were included in the analyses only if the prevoid total bladder volume (assessed by ultrasound) was ≥150 to ≤550 mL and the voided volume (V-comp) was >=125 mL.
Time Frame: Baseline, 12 weeks
Population: as for outcome 14
Measure: Median (Standard Deviation); unit: milliliters per second (mL/sec)
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 147 | 156 | 145
milliliters per second (mL/sec) | 0.10 (2.72) [-0.90 to 1.80] | 1.25 (3.24) [-0.30 to 3.25] | 0.70 (3.03) [-0.40 to 2.50]

16. Secondary Outcome: Change From Baseline in Volume of Voided Urine (V-Comp) at 12 Weeks
Description: V-comp (volume of urine voided) was measured in milliliters (mL) using a standard calibrated flowmeter. At each visit, a uroflowmetry assessment was considered valid and data were included in the analyses only if the prevoid total bladder volume (assessed by ultrasound) was ≥150 to ≤550 mL and V-comp was ≥125 mL.
Time Frame: Baseline, 12 weeks
Population: as for outcome 14
Measure: Median (Standard Deviation); unit: milliliter (mL)
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 147 | 156 | 145
milliliter (mL) | 0.0 (110.92) [-61.00 to 69.00] | 11.0 (101.45) [-64.00 to 70.50] | 16.0 (109.30) [-38.00 to 79.00]

17. Secondary Outcome: Change From Baseline in Postvoid Residual Volume (PVR) at 12 Weeks
Description: PVR was the amount of urine remaining in the bladder after void completion.
Time Frame: Baseline, 12 weeks
Population: as for outcome 14
Measure: Median (Standard Deviation); unit: milliliter (mL)
Arm/Group | Placebo | Tadalafil 5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 157 | 163 | 156
milliliter (mL) | 0.0 (56.48) [-20.0 to 23.0] | -1.0 (46.97) [-28.0 to 18.0] | -5.5 (59.21) [-23.5 to 17.0]
Statistical Analysis 1: Comparison: Placebo vs Tadalafil 5 mg; Test type: Superiority or Other; p = 0.303, ANOVA — [p-value comment as in outcome 14, analysis 1]; Analysis of variance (ANOVA) using rank transformed data
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.146, ANOVA — [p-value comment as in outcome 14, analysis 2]; ANOVA using rank transformed data

ADVERSE EVENTS:
Arm/Group | Tadalafil 5 mg | Tamsulosin 0.4 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/171 | 2/168 | 0/172
Other Adverse Events (participants affected / at risk) | 39/171 | 40/168 | 35/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil 5 mg (N=171) | Tamsulosin 0.4 mg (N=168) | Placebo (N=172)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil 5 mg (N=171) | Tamsulosin 0.4 mg (N=168) | Placebo (N=172)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3) | 8 (8)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Semen volume decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0)
Sebaceous adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 5 (5) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 6 (7) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 1 (4) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Retrograde ejaculation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Meniscus removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days